CLINICAL TRIAL: NCT05205616
Title: In-person Randomized Control Trial of the Incidence of Postoperative Hypoesthesia Among Bilateral Sagittal Split Osteotomy Patients Treated With Ultrasonic vs. Reciprocating Saw Instrumentation
Brief Title: Trial of Bilateral Sagittal Split Osteotomy Induced Paresthesia Using Ultrasonic vs. Reciprocating Saw Instrumentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21-33674
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Surgical Complication; Paresthesia; Fracture; Nerve Injury; Nerve Entrapments; Mandibular Nerve Injuries; Mandibular Hypoplasia; Mandibular Retrognathism; Mandibular Hyperplasia; Mandibular Prognathism
Keywords: Paresthesia; BSSO; Bilateral Saggital Split Osteotomy; Unfavorable split; Unfavorable fracture; Inferior Alveolar Nerve; Reciprocating Saw; Ultrasonic Saw; Pair matched; Randomized Control Trial
MeSH Terms: conditions — Paresthesia; Fractures, Bone; Nerve Compression Syndromes; Mandibular Nerve Injuries; Micrognathism; Malocclusion, Angle Class III

STUDY DESIGN:
Intervention Model Description: A matched-pair (with-in person) RCT design will be used, wherein one mandibular side (right versus left) in each patient will be randomized to be treated with Sonopet ultrasonic device (with the remaining side being treated with reciprocating saw). Neurosensory impairment, as herein described, will be compared at various post-operative times for a total follow-up of 3 months for each patients. Patients and the researchers examining patients post-operatively will be blinded.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and providers assessing postoperative nerve functioning are blinded to which side of the mandible received which intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Reciprocating saw (Placebo Comparator): The traditional surgical instrument used for cutting bilateral sagittal split osteotomies
  Interventions: Device: Reciprocating saw
- Sonopet ultrasonic saw (Active Comparator): This instrument is being compared to the reciprocating saw
  Interventions: Device: Sonopet ultrasonic saw

INTERVENTIONS:
Device: Sonopet ultrasonic saw — Ultrasonic saw to be used on a randomized side of the mandible, reciprocating saw will be used on other side
  Arms: Sonopet ultrasonic saw
Device: Reciprocating saw — See above description
  Arms: Reciprocating saw

SUMMARY:
The aim of this prospective study is to analyze the postoperative paresthesias experienced in patients who undergo bilateral sagittal split osteotomies (BSSO) using an ultrasonic saw, versus a reciprocating saw. Patients included in the study are ages 15-45 scheduled to undergo BSSO surgery at the University of California, San Francisco. One side of the patient's mandible will be instrumented with either the Stryker Sonopet ultrasonic saw or traditional reciprocating saw, while the other side will receive the remaining intervention (determined via randomization on the day of surgery). Patient paresthesias will then be analyzed on each side for 3 months postoperatively (at postoperative days: 1, 7, 14, 28, and 84). Sensory examinations will be carried out by blinded examiners using von Frey hairs and two point discrimination testing. Patients will also subjectively rate their sensation on each side. The results will then be analyzed to determine if patient paresthesias, including the severity and duration, differed depending on which instrument was used, the ultrasonic or reciprocating saw.

ELIGIBILITY:
Inclusion Criteria:

* Must be undergoing bilateral sagittal split osteotomy surgery with Dr. Saghezchi at UCSF
* Must agree to return for all follow up visits.
* Must not have any preexisting V3 nerve paresthesia
* Must be below the age of 45.

Exclusion Criteria:

* Persons with preexisting V3 nerve paresthesias
* Pre-pubertal children will be excluded (per routine practice for this type of surgery).
* Patients with syndromic genetic conditions that demonstrate clearly different anatomy in the two sides of their jaws will be excluded since the two sides may not be "exchangeable".

Max Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sohail Saghezchi, DDS, MD, Principal Investigator — UC San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco Medical Center, San Francisco, California
  - UCSF Benioff Children's Hospital, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Please note that since this is a pair-matched "split-mouth" study, where each participant was in both arms of the study since their left and right mandibles were the units receiving the different interventions in the study. Therefore, the total persons enrolled was 32 persons, while the total mandibles enrolled was 64.
Units Other Than Participants: Mandibular Rami
Period: Overall Study
Arm/Group | Reciprocating Saw | Sonopet Ultrasonic Saw
Started (Each study participant was assigned to both study arms, while only one of their two mandibular rami was assigned to that study arm.) | 32; 32 Mandibular Rami | 32; 32 Mandibular Rami
Completed (Each study participant was assigned to both study arms, while only one of their two mandibular rami was assigned to that study arm.) | 28; 28 Mandibular Rami | 28; 28 Mandibular Rami
Not Completed | 4; 4 Mandibular Rami | 4; 4 Mandibular Rami
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Population: Each study participant was assigned to both study arms, while only one of their two mandibular rami was assigned to that study arm, and received that treatment. Since 4 persons were lost to followup, the baseline participants groups only contains 28 persons.
Units Other Than Participants: Mandibular Rami
Groups:
- Total: Total of all reporting groups
Arm/Group | Reciprocating Saw | Sonopet Ultrasonic Saw | Total
Number analyzed (Participants) | 28 | 28 | 28
Number analyzed (Mandibular Rami) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] — Please note that this is a "split-mouth" study, where each participant is enrolled in both arms of the study.
  years | 25.95 (9.8) | 25.95 (9.8) | 25.95 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 13 | 13 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 13 | 13 | 26
  African American | 1 | 1 | 2
  Latinx | 8 | 8 | 16
  Asian | 6 | 6 | 12
Normal Baseline VFH Score (Lightest VFH Filament sensed has a weight of 0.008g) [Count of Units; unit: Mandibular Rami] — VFH filaments are used to measure the lightest force sensed by a dermatome in question. In this study, the measurements range from: 0.008g, 0.02g, 0.04g, 0.07g, 0.16g, 0.4g, 0.6g, 1g, 1.4g, 2g, 4g, 6g, 8g, 10g, 15g. Someone who can sense the finest measurement of 0.008g is said to have no neurosensory deficit, hence a "Normal Baseline VFH Score".
  Mandibular Rami | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Hypoesthesia Experienced at 3months
Description: Count of patient mandibles who exhibited **any** hypoesthesia at 3months post-operation (i.e. VFH does not equal 0.008g). VFH filaments measure the minimum weight which a dermatome in question can sense. In this study, the measurements were designed to have the following range: 0.008g, 0.02g, 0.04g, 0.07g, 0.16g, 0.4g, 0.6g, 1g, 1.4g, 2g, 4g, 6g, 8g, 10g, 15g, with 0.008g being no neurosensory deficit. Although 28 persons completed the study, only 21 patients presented for their 3 month followup time, which was defined as with-in 15 days of 90th day after operation. Therefore, the denominator for this outcome is 21, for each intervention arm. The numerator is the number of Left or Right chin areas that exhibited less than "normal" sensation.
Time Frame: Within 15 days of exact 3 months post-operation
Population: Although 28 persons completed the study, only 21 patients presented for their 3 month followup time, which was defined as with-in 15 days of 90th day after operation.
Measure: Count of Units; unit: Left or Right Chin Area
Units Other Than Participants: Left or Right Chin Area
Arm/Group | Reciprocating Saw | Sonopet Ultrasonic Saw
Number analyzed (Participants) | 21 | 21
Number analyzed (Left or Right Chin Area) | 21 | 21
Left or Right Chin Area | 8 | 3

2. Secondary Outcome: Unfavorable Fracture
Description: When a saggital split osteotomy is performed, a controlled fracture of the mandibular ramus is induced which follows an exact intended path of fracture. An unfavorable fracture is one that does not follow this exact path of fracture, and needs to be surgically mended. An unfavorable fracture is associated with poorer post-operative recovery.
Time Frame: This outcome occurs during the surgery. It was measured on the same day.
Population: Each study participant was enrolled in both study arms, but only one of each person's two mandible was randomized to each study arm.
Measure: Count of Units; unit: Mandibular rami
Units Other Than Participants: Mandibular rami
Arm/Group | Reciprocating Saw | Sonopet Ultrasonic Saw
Number analyzed (Participants) | 28 | 28
Number analyzed (Mandibular rami) | 28 | 28
Mandibular rami | 2 | 0

ADVERSE EVENTS:
Time Frame: At a minimum each participant who was not lost to follow up was followed for three months (defined as 85 - 115 days) after their operation. However, patients were followed as long as they return for assessment of their orthognathic surgery. The follow up of participants who completed the study ranged from 85 days to 419 days.
Arm/Group | Reciprocating Saw | Sonopet Ultrasonic Saw
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 4/28 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reciprocating Saw (N=28) | Sonopet Ultrasonic Saw (N=28)
Transaction of Inferior Alveolar Nerve (IAN), which provides sensation to the chin area (Surgical and medical procedures) | 4 (4) | 1 (1) — This study tested the effect of using two different kinds of cutting saws on neurosensory outcomes of the left or right chin areas. The sensation to this area is provided by the IAN, which is always at risk of being transacted during this surgery.

LIMITATIONS AND CAVEATS:
Given the relatively few secondary outcome occurrences, unfavorable mandibular fractures, which occurred in 2/28 in the reciprocating saw arm and 0/28 in the ultrasonic saw arm, it is not possible to meaningfully interpret the findings for the secondary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT05205616/Prot_SAP_003.pdf